CLINICAL TRIAL: NCT01592851
Title: A Clinical Study Investigating the Efficacy of a Dentifrice in Providing Short Term Relief From Dentinal Hypersensitivity
Brief Title: Clinical Efficacy of a Toothpaste in Providing Relief From the Pain of Dentinal Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RH01324
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-02

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Dentifrice containing stannous fluoride
  Interventions: Drug: Stannous Fluoride
- Arm 2 (Active Comparator): Marketed dentifrice containing Sodium Monofluorophosphate
  Interventions: Drug: Sodium Monofluorophosphate

INTERVENTIONS:
Drug: Stannous Fluoride — dentifrice containing stannous fluoride
  Arms: Arm 1
Drug: Sodium Monofluorophosphate — dentifrice containing Sodium Monofluorophosphate
  Arms: Arm 2

SUMMARY:
A study to compare the efficacy of a test dentifrice against a control dentifrice in reducing dentinal hypersensitivity over a two week treatment period.

ELIGIBILITY:
- Subjects who suffer from tooth sensitivity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- BioSci Research America, Inc., Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Parkinson CR, Hughes N, Hall C, Whelton H, Gallob J, Mason S. Three randomized clinical trials to assess the short-term efficacy of anhydrous 0.454% w/w stannous fluoride dentifrices for the relief of dentin hypersensitivity. Am J Dent. 2016 Feb;29(1):25-32. PMID 27093773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 126 participants screened, 9 participants did not meet the study criteria, 3 were lost to follow up and 1 withdrew consent before randomization. Remaining 113 participants were randomized to study treatments.
Groups:
- Stannous Fluoride (SnF) Dentifrice: Participants brushed each of the 2 selected sensitive teeth for 30 seconds each, followed by the whole mouth with 1 inch strip of the test dentifrice (0.454% SnF) for at least 1 minute and rinsing with 5mL of water.
- Sodium Monofluorophosphate (NaMFP) Dentifrice: Participants brushed whole mouth with 1-inch strip of the control dentifrice (0.76% Sodium Monofluorophosphate [NaMFP]) for one timed minute, followed by rinsing with 5 mL of water.
Period: Overall Study
Arm/Group | Stannous Fluoride (SnF) Dentifrice | Sodium Monofluorophosphate (NaMFP) Dentifrice
Started | 56 | 57
Completed | 56 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SnF Dentifrice: Participants brushed each of the 2 selected sensitive teeth for 30 seconds each, followed by the whole mouth with 1 inch strip of the test dentifrice (0.454% SnF) for at least 1 minute and rinsing with 5mL of water.
- NaMFP Dentifrice: Participants brushed whole mouth with 1-inch strip of the control dentifrice (0.76% NaMFP) for one timed minute, followed by rinsing with 5 mL of water.
- Total: Total of all reporting groups
Arm/Group | SnF Dentifrice | NaMFP Dentifrice | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (10.70) | 34.8 (9.86) | 36.5 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 79
  Male | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Evaporative Air Sensitivity Pain Response on a Schiff Sensitivity Scale at Day 14
Description: Response to a constant jet of air applied to hypersensitive teeth is evaluated using a Schiff Sensitivity pain response scale. According to this analog scale, pain response for each individual stimulated tooth ranged from 0 to 3; 0 - participant does not respond to air stimulation, 1 - participant responds to air stimulus but does not request discontinuation of stimulus, 2 - participant responds to air stimulus and request discontinuation of stimulus, 3 - participant responds to air stimulus, considers stimulus to be painful and request discontinuation of stimulus. Those teeth that met the tactile threshold inclusion criterion (tactile threshold ≤ 20g) were assessed at baseline and Day 14. The Investigator directed a second application of air from a standard dental syringe to the facial surface of the two sensitive teeth selected at baseline. The Schiff Sensitivity Score was calculated as the subject level mean change (on two teeth) from baseline.
Time Frame: Baseline to Day 14
Population: Intent To Treat (ITT) population: All randomized participants, who were administered with at least one study treatment during the study and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 56 | 57
Score on a scale | -1.20 (0.70) | -0.37 (0.43)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = -0.83, 95% CI 2-sided [-1.03 to -0.63] — Difference is 0.454% SnF minus 0.76% NaMFP such that a negative difference favours first named treatment

2. Secondary Outcome: Change From Baseline in Evaporative Air Sensitivity Pain Response on a Schiff Sensitivity Scale Immediately Post-treatment
Description: Response to a constant jet of air applied to hypersensitive teeth is evaluated using a Schiff Sensitivity pain response scale. According to this analog scale, pain response for each individual stimulated tooth ranged from 0 to 3; 0 - participant does not respond to air stimulation, 1 - participant responds to air stimulus but does not request discontinuation of stimulus, 2 - participant responds to air stimulus and request discontinuation of stimulus, 3 - participant responds to air stimulus, considers stimulus to be painful and request discontinuation of stimulus. Those teeth that met the tactile threshold inclusion criterion (tactile threshold ≤ 20g) were assessed at baseline and immediately after treatment. The Investigator directed a second application of air from a standard dental syringe to the facial surface of the two sensitive teeth selected at baseline. The Schiff Sensitivity Score was calculated as the subject level mean change (on two teeth) from baseline.
Time Frame: Baseline to immediately post treatment administration
Population: ITT population: All randomized participants, who were administered with at least one study treatment during the study and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 56 | 57
Score on a scale | -0.40 (0.46) | -0.14 (0.35)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p = 0.0006, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = -0.26, 95% CI 2-sided [-0.41 to -0.12] — Difference is 0.454% SnF minus 0.76% NaMFP such that a negative difference favours first named treatment

3. Secondary Outcome: Change From Baseline in Evaporative Air Sensitivity Pain Response on a Schiff Sensitivity Scale at Day 3
Description: Response to a constant jet of air applied to hypersensitive teeth is evaluated using a Schiff Sensitivity pain response scale. According to this analog scale, pain response for each individual stimulated tooth ranged from 0 to 3; 0 - participant does not respond to air stimulation, 1 - participant responds to air stimulus but does not request discontinuation of stimulus, 2 - participant responds to air stimulus and request discontinuation of stimulus, 3 - participant responds to air stimulus, considers stimulus to be painful and request discontinuation of stimulus. Those teeth that met the tactile threshold inclusion criterion (tactile threshold ≤ 20g) were assessed at baseline and Day 3. The Investigator directed a second application of air from a standard dental syringe to the facial surface of the two sensitive teeth selected at baseline. The Schiff Sensitivity Score was calculated as the subject level mean change (on two teeth) from baseline.
Time Frame: Baseline to Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 56 | 57
Score on a scale | -0.70 (0.60) | -0.25 (0.39)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = -0.45, 95% CI 2-sided [-0.63 to -0.28] — Difference is 0.454% SnF minus 0.76% NaMFP such that a negative difference favours first named treatment

4. Secondary Outcome: Change From Baseline in Tactile Pain Threshold Score at Day 14
Description: The Response to increasing force on hypersensitive teeth was evaluated using a Yeaple Probe pain response scale (10g to 80g). According to this tactile sensitivity assessment, an increasing force is applied to hypersensitive tooth until a yes response to pain is recorded or the maximum force has been reached. Tactile testing begins with a force of 10g and it is increased by 10g, with each successive challenge, until either a "yes" response is recorded or the maximum force (80g) is reached. An increase in tactile score from baseline represents an improvement in sensitivity
Time Frame: Baseline to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Force (grams)
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 56 | 57
Force (grams) | 22.9 (21.14) | 3.5 (5.67)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = 19.42, 95% CI 2-sided [13.70 to 25.15] — Difference is 0.454% SnF minus 0.76% NaMFP such that a positive difference favours first named treatment

5. Secondary Outcome: Change From Baseline in Tactile Pain Threshold Score at Day 3
Description: as for outcome 4
Time Frame: Baseline to Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Force (grams)
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 56 | 57
Force (grams) | 9.8 (15.52) | 3.0 (4.90)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p = 0.0021, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = 6.84, 95% CI 2-sided [2.54 to 11.13] — Difference is 0.454% SnF minus 0.76% NaMFP such that a positive difference favours first named treatment

6. Secondary Outcome: Change From Baseline in Tactile Pain Threshold Score Immediately Post-treatment
Description: as for outcome 4
Time Frame: Baseline to immediately post treatment administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Force (grams)
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 56 | 57
Force (grams) | 5.8 (10.17) | 1.9 (3.24)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p = 0.0070, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean DIfference = 3.87, 95% CI 2-sided [1.08 to 6.65] — Difference is 0.454% SnF minus 0.76% NaMFP such that a positive difference favours first named treatment

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product, or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/57
Other Adverse Events (participants affected / at risk) | 0/56 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.